CLINICAL TRIAL: NCT02548026
Title: Meals and Grazing Study
Acronym: MAGS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 7439
Record Dates: First submitted 2015-09-08; First posted 2015-09-14 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-09

CONDITIONS: Healthy
Keywords: meal frequency; eating frequency; ingestive frequency; positive energy balance; satiety; appetite; hunger

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Eating Frequency (High EF) (Experimental): 8 Eating Occasions
  Interventions: Behavioral: High Eating Frequency (High EF)
- Low Eating Frequency (High EF) (Experimental): 3 Eating Occasions
  Interventions: Behavioral: Low Eating Frequency (Low EF)

INTERVENTIONS:
Behavioral: High Eating Frequency (High EF) — Free-living participants complete a 21-day high eating frequency (high EF) Phase in which they consume all daily energy at 8 eating occasions.
  Arms: High Eating Frequency (High EF)
Behavioral: Low Eating Frequency (Low EF) — Free-living participants complete a 21-day low eating frequency (low EF) Phase in which they consume all daily energy at 3 eating occasions.
  Arms: Low Eating Frequency (High EF)

SUMMARY:
The purpose of this study was to determine the effects of low vs. high eating frequency (EF) on biomarkers of health and subjective appetite.

DETAILED DESCRIPTION:
Observational studies have demonstrated an inverse relationship between eating frequency (EF), obesity, and other markers for disease risk. It has been suggested that consumption of several small, frequent meals may influence physiological mechanisms, reducing the risk for disease and lowering appetite. Participants in this randomized crossover study completed two intervention phases lasting three weeks each: one of low eating frequency ("low-EF"; 3 eating occasions/day) and one of high eating frequency ("high-EF"; 8 eating occasions/day). Fasting C-reactive protein, insulin-like growth factor, and leptin were measured at baseline and endpoint of each phase and an optional subjective appetite testing session lasting four hours was offered at the endpoint of each phase. During appetite testing sessions, participants consumed an amount of food equal in total energy and macronutrient content at either one occasion at 8:00 am ("low-EF" condition) or spread evenly over two smaller eating occasions at 8:00 am and 10:30 am ("high-EF" condition). Ratings of hunger, desire to eat, fullness, thirst, and nausea were made every 30 minutes using paper-and-pencil semi-anchored 100-mm Visual Analog Scales. A composite appetite score was calculated as the mean of hunger, desire to eat, and 100-fullness. The generalized estimating equation modification of linear regression was used to compare fasting plasma biomarkers and mean ratings of subjective appetite.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be overweight and obese (BMI 25 and over) males and females ages 18-50 years.
* Participants must be willing to report to FHCRC on 5 occasions (initial screening appointment + 4 testing sessions)
* Participants must be willing to provide a 7-day food record for analysis prior to Phase 1 and Phase 2 of the study
* Participants must be willing to follow diet protocol during Phase 1 of the study
* Participants must be willing to undergo 4 blood draws

Exclusion Criteria:

* Non-diabetic (self-report)
* Non-smokers (self-report)
* Not following a diet to gain or lose weight (self-report)
* Normal cholesterol (self-report)
* Normal blood pressure (self-report)
* Not currently taking any medication (self-report)
* Not pregnant or nursing (self-report and verification by DEXA)
* Not athletes in training (self-report)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2011-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Inflammatory biomarkers in high vs. low eating frequency conditions | 3 weeks
  Inflammatory biomarkers in high vs. low eating frequency conditions

SECONDARY OUTCOMES:
Subjective appetite in high vs. low eating frequency conditions | 4 hours
  Subjective appetite as reported using visual analog scale in high vs. low eating frequency conditions

CONTACTS AND LOCATIONS:
Overall Officials: Marian Neuhouser, PhD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Perrigue MM, Drewnowski A, Wang CY, Neuhouser ML. Higher Eating Frequency Does Not Decrease Appetite in Healthy Adults. J Nutr. 2016 Jan;146(1):59-64. doi: 10.3945/jn.115.216978. Epub 2015 Nov 11. PMID 26561409